CLINICAL TRIAL: NCT02447029
Title: Self-Administered Lidocaine Gel for Pain Management With First Trimester Surgical Abortion: A Randomized Controlled Trial
Acronym: SALSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vaginal Lidocaine
Record Dates: First submitted 2014-12-01; First posted 2015-05-18 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy, Unwanted
Keywords: abortion; pain management
MeSH Terms: conditions — Agnosia | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Comparator (Experimental): Drug: vaginal 2% Xylocaine
  Interventions: Drug: vaginal 2% Xylocaine
- standard lidocaine paracervical block (Other): standard lidocaine paracervical block
  Interventions: Drug: standard lidocaine paracervical block

INTERVENTIONS:
Drug: vaginal 2% Xylocaine — patient-administered vaginal lidocaine jelly versus provider-administered standard lidocaine paracervical block
  Arms: Active Comparator
Drug: standard lidocaine paracervical block — 1% lidocaine paracervical injection
  Arms: standard lidocaine paracervical block

SUMMARY:
Despite global efforts to decrease discomfort during surgical abortion, pain remains a limiting factor in where and how procedures are performed. Several studies have investigated different methods of delivering cervical anesthesia prior to abortion, however to the best of the investigators' knowledge, there is no published data that 1) rigorously examines the effect of a time interval between local anesthetic administration and procedure initiation, or 2) explores whether adequate pain relief is possible through self-administered, non-invasive means alone. Research in this area has a significant public health impact, given the large number of women worldwide who seek abortions.

The investigators propose to explore the effect of a locally applied vaginal lidocaine gel in place of the traditional paracervical block prior to first trimester surgical abortion. They hypothesize that lidocaine gel is no worse than paracervical block at decreasing abortion related pain at a variety of time points throughout the procedure. This is a non-inferiority, open label, randomized controlled trial.

If self-administered vaginal gel is acceptable and effective, it would increase options for pain control during abortion and other gynecologic procedures.

DETAILED DESCRIPTION:
Abortion remains one of the most common surgical procedures in the world, regardless of region or development status [Guttmacher 2012]. In the United States, at least half of all women will experience an unintended pregnancy by age 45, and one third of all women will have had an abortion by this same age [Guttmacher 2014].

Despite universal efforts to increase the comfort of these procedures, pain remains a limiting factor in where and how abortion is performed. Recent estimates reveal that 70-97% of women experience pain during abortion [Renner 2010, Paul 2009, Belanger 1988]. Strategies to reduce all aspects of abortion related pain have the potential for significant public health impact, given the large number of women who seek these services. A survey of National Abortion Federation clinics found that to date, most providers (84%) employ the use of a lidocaine paracervical block for cervical anesthesia prior to abortion [O'Connell 2009], but traditionally without a waiting period between lidocaine administration and procedure initiation.

To the best of our knowledge, there are no published studies that 1) rigorously examine the effect of a time interval between local anesthetic administration and procedure initiation, or 2) explore whether adequate pain relief is possible through self-administered, non-invasive means alone. The investigators propose to explore the effect of a locally applied lidocaine gel in place of the traditional paracervical block to decrease abortion related pain.

The objective of this study is to compare pain control at various time points during first trimester surgical abortion using a locally applied, patient-administered lidocaine gel as compared to traditional lidocaine paracervical block.

If a patient-administered vaginal gel is acceptable and effective, it would increase options for pain control during abortion and other gynecologic procedures, and perhaps replace paracervical injection altogether.

Hypothesis: Patients who receive lidocaine gel applied 30 minutes prior to first trimester surgical abortion will have pain control equivalent to that of a traditional paracervical block.

This is a non-inferiority, open-label, randomized controlled trial of women ages 18 and older undergoing first trimester surgical abortion at 50/7 to 116/7 weeks.

ELIGIBILITY:
Inclusion criteria:

* Women ages 18 and older undergoing elective surgical abortion at 5 and 0/7 to 11 and 6/7 weeks gestational age
* Use of IV sedation for pain management
* English or Spanish speaking
* Ability to give informed consent

Exclusion criteria:

* Any pre-operative use of misoprostol (typically given at 12 weeks and above in this clinic)
* Allergy to study medications: lidocaine, midazolam, fentanyl
* Known uterine anomaly
* Prior cervical surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Planned Parenthood Mar Monte, San Jose, California, United States

REFERENCES:
- [Derived] Conti JA, Lerma K, Shaw KA, Blumenthal PD. Self-Administered Lidocaine Gel for Pain Control With First-Trimester Surgical Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2016 Aug;128(2):297-303. doi: 10.1097/AOG.0000000000001532. PMID 27400015

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Comparator | Standard Lidocaine Paracervical Block
Started | 72 | 70
Treated | 69 | 68
Completed | 69 | 68
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: Treated participants were analyzed for baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator | Standard Lidocaine Paracervical Block | Total
Number analyzed (Participants) | 69 | 68 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 69 | 68 | 137
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 68 | 137
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Difference in Pain Level at Time of Cervical Dilation as Measured by a Visual Analog Scale
Description: This is the amount of pain self-reported by the patient at the time of cervical dilation. VAS ranged from 0 to 100 mm, 0 equals no pain, 100 equals worse pain imaginable.
Time Frame: At time of cervical dilation, 30 minutes after lidocaine administration
Population: Treated participants were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active Comparator | Standard Lidocaine Paracervical Block
Number analyzed (Participants) | 69 | 68
units on a scale | 68 [17 to 97] | 65 [10 to 100]

2. Secondary Outcome: Pain Level Prior to Procedure (Anticipated Pain) as Measured by a Visual Analog Scale
Description: This is the amount of pain self-reported by the patient prior to the procedure (Anticipated pain). VAS ranged from 0 to 100 mm, 0 equals no pain, 100 equals worse pain imaginable.
Time Frame: Pain level prior to procedure
Population: Treated patients were included in the analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active Comparator | Standard Lidocaine Paracervical Block
Number analyzed (Participants) | 69 | 68
units on a scale | 59 [3 to 98] | 56 [12 to 99]

3. Secondary Outcome: Pain With Speculum Insertion as Measured by a Visual Analog Scale
Description: This is the amount of pain self-reported by the patient at the time of speculum insertion. VAS ranged from 0 to 100 mm, 0 equals no pain, 100 equals worse pain imaginable.
Time Frame: Pain at time of speculum insertion
Population: Treated patients were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator | Standard Lidocaine Paracervical Block
Number analyzed (Participants) | 69 | 68
units on a scale | 19.5 (18.4) | 22.3 (19.5)

4. Secondary Outcome: Pain With Tenaculum Placement as Measured by a Visual Analog Scale
Description: This is the amount of pain self-reported by the patient at the time of tenaculum placement. VAS ranged from 0 to 100 mm, 0 equals no pain, 100 equals worse pain imaginable.
Time Frame: Pain at time of tenaculum placement
Population: All treated patients were included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Comparator | Standard Lidocaine Paracervical Block
Number analyzed (Participants) | 69 | 68
units on a scale | 39.8 (22.3) | 32.4 (24.3)

5. Secondary Outcome: Pain 30-45 Minutes After Procedure as Measured by a Visual Analog Scale
Description: This is the amount of pain self-reported by the patient 30-45 minutes after procedure. VAS ranged from 0 to 100 mm, 0 equals no pain, 100 equals worse pain imaginable.
Time Frame: Pain prior to discharge home: 30-45 minutes after completion of procedure
Population: All treated patients were included in the analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active Comparator | Standard Lidocaine Paracervical Block
Number analyzed (Participants) | 69 | 68
units on a scale | 9 [0 to 85] | 11.5 [0 to 90]

6. Secondary Outcome: Overall Satisfaction With Procedure as Measured by a Visual Analog Scale
Description: This is the level of overall satisfaction self-reported by the patient at the completion of the procedure and prior to discharge. VAS ranged from 0 to 100 mm, 0 equals not satisfied, 100 equals highest satisfaction possible.
Time Frame: 30-45 minutes after completion of procedure
Population: All treated patients were included in the analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active Comparator | Standard Lidocaine Paracervical Block
Number analyzed (Participants) | 69 | 68
units on a scale | 86 [0 to 99] | 92.5 [44 to 100]

7. Secondary Outcome: Overall Complication Rate as Measured by a Count of Participants in Each Group
Time Frame: Rate of complications at the end of the study
Population: All treated patients were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator | Standard Lidocaine Paracervical Block
Number analyzed (Participants) | 69 | 68
Participants | 0 | 0

ADVERSE EVENTS:
Description: Treated participants were included in the analysis.
Arm/Group | Active Comparator | Standard Lidocaine Paracervical Block
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/68
Other Adverse Events (participants affected / at risk) | 0/69 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No